CLINICAL TRIAL: NCT02168075
Title: Can Mannitol Increments Provide More Brain Relaxation in Patients Undergoing Craniotomy for Supratentorial Brain Tumor Removal?
Brief Title: Mannitol Brain Relaxation Effect
Acronym: MANNITOL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hee-Pyoung Park, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Mannitol
Record Dates: First submitted 2014-06-16; First posted 2014-06-20 (Estimated); Last update posted 2014-10-24 (Estimated); Status verified 2014-10

CONDITIONS: Supratentorial Neoplasms
MeSH Terms: conditions — Supratentorial Neoplasms | interventions — Mannitol

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group 1 (Experimental): 0.25g/kgof 20% mannitol administered at drilling of skull.
  Interventions: Drug: 0.25g/kgof 20% mannitol
- Group 2 (Experimental): 0.5g/kg of 20% mannitol administered at drilling of skull.
  Interventions: Drug: 0.5g/kg of 20% mannitol
- Group 3 (Experimental): 1.0 g/kg of 20% mannitol administered at drilling of skull.
  Interventions: Drug: 1.0g/kg of 20% mannitol
- Group 4 (Experimental): 1.5g/kg of 20% mannitol administered at drilling of skull.
  Interventions: Drug: 1.5g/kg of 20% mannitol

INTERVENTIONS:
Drug: 0.25g/kgof 20% mannitol — When the neurosurgeon starts the drilling of skull, 0.25g/kg of 20% mannitol administered through the IV catheter with fulldrip. Neurosurgeon evaluate the degree of brain relaxation after dura opening in 4 point scale ( 1=bulging brain, 2=firm brain, 3-satisfactorily relaxed, 4=perfectly relaxed).
  Arms: Group 1
Drug: 0.5g/kg of 20% mannitol — When the neurosurgeon starts the drilling of skull, 0.5g/kg of 20% mannitol administered through the IV catheter with fulldrip. Neurosurgeon evaluate the degree of brain relaxation after dura opening in 4 point scale ( 1=bulging brain, 2=firm brain, 3-satisfactorily relaxed, 4=perfectly relaxed).
  Arms: Group 2
Drug: 1.0g/kg of 20% mannitol — When the neurosurgeon starts the drilling of skull, 1.0g/kg of 20% mannitol administered through the IV catheter with fulldrip. Neurosurgeon evaluate the degree of brain relaxation after dura opening in 4 point scale ( 1=bulging brain, 2=firm brain, 3-satisfactorily relaxed, 4=perfectly relaxed).
  Arms: Group 3
Drug: 1.5g/kg of 20% mannitol — When the neurosurgeon starts the drilling of skull,1.5g/kg of 20% mannitol administered through the IV catheter with fulldrip. Neurosurgeon evaluate the degree of brain relaxation after dura opening in 4 point scale ( 1=bulging brain, 2=firm brain, 3-satisfactorily relaxed, 4=perfectly relaxed).
  Arms: Group 4

SUMMARY:
Mannitol is widely used in patients with elevated intracranial pressure. In neurosurgical field, especially in large size or with brain edema, it is necessary to decrease brain volume to facilitate surgical approach. In general, 0.25 -1.5g of mannitol per kilogram has been known to decrease ICP effectively. But there are some debates in regard to appropriate dose of mannitol.

DETAILED DESCRIPTION:
Previous meta-analysis reported that mannitol has dose-response relationship with intracranial pressure. Another study of Sorani showed dose-response relationship between mannitol and intracranial pressure (ICP) in traumatic brain injury patients.

In this study, authors would investigate that mannitol increments can provide more brain relaxation in patients undergoing craniotomy for supratentorial brain tumor removal.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent craniotomy for supratentorial brain tumor under general anesthesia

Exclusion Criteria:

* Patient who does not agree to the study
* Patients with or American Society of Anesthesiologists (ASA) physical status class IV or more
* Patients with glasgow coma scale (GCS) under 13 points
* Patients who have hyponatremia or hypernatremia (Na<130 or >150mEq/L)
* Patients who have congestive heart failure or moderately decreased renal function (GFR <60ml/min/1.73m2)
* Patients with extraventricular drainage such as external ventricular drain (EVD) or ventriculoperitoneal (VP) shunt
* Patients who already under mannitolization

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2014-06; Primary Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
brain parenchymal relaxation | intraoperative
  Brain relaxation was assessed immediately after opening of the dura on a scale range from 1 to 4 (1=bulging brain, 2=firm brain, 3-satisfactorily relaxed, 4=perfectly relaxed) by neurosurgeon who is blinded to dose of mannitol.
  3 and 4 scale means brain relaxed. We would analyse if the success proportion of brain relaxation increase according to the mannitol increment 0.25g/kg, 0.5g/kg, 1.0g/kg and 1.5g/kg using Cochran-Armitage trend test.

SECONDARY OUTCOMES:
Hemodynamic change | at baseline, 30 min, 60min and 180 min after the administration of the study drug
  Check the mean arterial blood pressure (ABP), heart rate (HR), central venous pressure (CVP) at baseline, 30min, 60min, and 180 min after skin incision. Baseline value means data of just after anesthetic induction.
Electrolyte change | at baseline, 30 min, 60min and 180 min after the administration of the study drug
  Check the serum laboratory result of electrolyte include potassium, sodium immediately before the infusion of mannitol and 30, 60 and 180 min after the administration of the study drug.
Brain relaxation score | intraoperative
  Brain relaxation was assessed immediately after opening of the dura on a scale range from 1 to 4 (1=bulging brain, 2=firm brain, 3-satisfactorily relaxed, 4=perfectly relaxed) by neurosurgeon who is blinded to dose of mannitol.
Urine output | at just after induction of anesthesia, 30min, 60min and 180 min after mannitl loading
  check the urine amount at baseline (just after induction of anesthesia), 30min/60min/180min after mannitol loading.
Osmolar gap change | at baseline, 30min, 60min and 180 min after the administration of the study drug
  Check the serum osmolarity, blood urea nitrogen (BUN), glucose immediately before the infusion of mannitol and 30, 60, and 180 minutes after the administration of the study drug for calculate the osmolar gap.
  Osmolar gap (OG) = measured osmolarity - calculated osmolarity Calculated osmolarity = 2x[Na(mMol)]+1.15x([glucose(mg/dL)/18)+([urea(mg/dL)/2.8)

OTHER OUTCOMES:
Arterial blood gas analysis (ABGA) change | at baseline, 30min, 60min and 180 min after the administration of the study drug
  Check the arterial blood gas analysis include (pH, PaCO2, PaO2, lactate and hematocrit) immediately before the infusion of mannitol and 30, 60, and 180 minutes after the administration of the study drug.

CONTACTS AND LOCATIONS:
Overall Officials: Hee Pyung Park, MD PhD, Study Director — Professor; Eugene Kim, MD, Principal Investigator — Clinical Instuctor
Locations (1):
- Seoul National University of Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Seo H, Kim E, Jung H, Lim YJ, Kim JW, Park CK, Se YB, Jeon YT, Hwang JW, Park HP. A prospective randomized trial of the optimal dose of mannitol for intraoperative brain relaxation in patients undergoing craniotomy for supratentorial brain tumor resection. J Neurosurg. 2017 Jun;126(6):1839-1846. doi: 10.3171/2016.6.JNS16537. Epub 2016 Aug 19. PMID 27540904